CLINICAL TRIAL: NCT05508269
Title: Quantitative Polymerase Chain Reaction of Four Genes in Coronary Artery Disease, Myocardial Infarction and Ischemic Cardiomyopathy
Brief Title: Genetics of Ischemic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Wageh Mohareb, PhD Mina Wageh Mohareb, Clinical researcher, Faculty of Pharmacy, Cairo University, Cairo University
Other Study IDs: RHFCS1
Record Dates: First submitted 2019-09-13; First posted 2022-08-19 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Ischemic Cardiomyopathy; qrt-pcr
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cardiac tissue specimens and blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control subjects: control cases who were diagonosed as healthy subjects after diagnostic catheterization
  Interventions: Genetic: quantitative polymerase chain reaction(QPCR) for four genes; Procedure: Cardiac biopsy, blood sampling
- Stable coronary artery disease: patients with stable coronary artery disease undergoing elective PCI who were diagnozed with coronary lesion/s and underwent stent implantation without previous history of myocardial infarction
  Interventions: Genetic: quantitative polymerase chain reaction(QPCR) for four genes; Procedure: Cardiac biopsy, blood sampling
- Myocardial infarction patients: patients with history of myocardial infarction or with acute myocardial infarction undergoing primary PCI
  Interventions: Genetic: quantitative polymerase chain reaction(QPCR) for four genes; Procedure: Cardiac biopsy, blood sampling
- Ischaemic cardiomyopathy patients: patients with ischaemic cardiomyopathy diagnosed by ejection fraction less than 35% with history of coronary artery disease or myocardial infarction or those with acute myocardial infarction with reduced ejection fraction.
  Interventions: Genetic: quantitative polymerase chain reaction(QPCR) for four genes; Procedure: Cardiac biopsy, blood sampling

INTERVENTIONS:
Genetic: quantitative polymerase chain reaction(QPCR) for four genes — quantitative polymerase chain reaction(QPCR) for four genes
Procedure: Cardiac biopsy, blood sampling — In the studied thirteen peripheral blood subjects, five milliliters blood samples were taken from each patient in potassium EDTA tubes, immediately inserted in liquid nitrogen container and then stored in -80 refrigerators. All studied thirteen cardiac tissue subjects were underwent cardiac biopsy after PCI in order to take two specimens from the left ventricle using judkin right seven french catheters for femoral access and cardiac bioptome 2.3 mm wide. All cardiac specimens were collected in cryotubes, immediately inserted in liquid nitrogen container and then stored in -80 refrigerators.

SUMMARY:
Background:Ischemic heart disease is one of the heaviest health-related burdens worldwide.We aimed to identify the common hub mRNA and pathways that are involved in pathological progression of ischemic cardiomyopathy. Methods: To explore potential differentially expressed genes (DEGs) of all ischemic heart disease stages, we used chipster and GEO2R tools to analyze of retrieved eight high throughput RNA datasets obtained from GEO database. Gene Ontology functional annotation and Pathways enrichment analyses were used to obtain the common functional enriched DEGs which were visualized in protein-protein interactions (PPI) network to explore the hub mRNA according to the interaction scores. Validation qRT-PCR was carried out for blood and cardiac biopsies compared with controls to validate the determined four hub mRNAs and subsequently reviewed inside comprehensive published meta-analysis database. The validated mRNAs were visualized in two interaction modules. Finally screening of approved drugs was applied.

ELIGIBILITY:
Inclusion criteria The enrolled patients aged 20-80 years with stable coronary artery disease undergoing elective PCI or patients with unstable angina or myocardial infarction undergoing rescue PCI and admitted to the cardiology hospital (Asyut University, Asyut, Egypt) were recruited in this study.

Exclusion criteria Patients with dilated cardiomyopathy were execluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects were categorized into three control cases who were diagonosed as healthy subjects after diagnostic catheterization, three patients with stable coronary artery disease undergoing elective PCI who were diagnozed with coronary lesion/s and underwent stent implantation without previous history of myocardial infarction, four patients with history of myocardial infarction or with acute myocardial infarction undergoing primary PCI and three patients with ischaemic cardiomyopathy diagnosed by ejection fraction less than 35% with history of coronary artery disease or myocardial infarction or those with acute myocardial infarction with reduced ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Genetic pathway of pathological progression from stable coronary artery disease to myocardial infarction and finally to ischaemic cardiomyopathy | 2 years
  The expected results may explain novel genetic pathways of the clinical progression of asymptomatic structural cardiac disorder (Stable coronary artery disease) to typically symptomatic ischaemic cardiomyopathy. Gene expression profiling of seven genes in RNA of all cardiac specimens was measured using QPCR analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- cardiology hospital (Asyut University, Asyut, Egypt), Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No